CLINICAL TRIAL: NCT00530855
Title: A Multicenter, Open-label Extension Trial to Assess the Long-term Use of Lacosamide Monotherapy and Safety of Lacosamide Monotherapy and Adjunctive Therapy in Subjects With Partial-onset Seizures
Brief Title: Trial to Assess Long-term Lacosamide (LCM) Monotherapy Use and Safety of LCM Monotherapy and Adjunctive Therapy for Partial-onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0904; 2007-005440-25 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2007-09-14; First posted 2007-09-18 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; Partial-onset Seizures; Lacosamide; Monotherapy; Vimpat
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

ARMS (1):
- Lacosamide (Experimental): Lacosamide tablets for dosing 100 -800 mg/day
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — 50 mg and 100 mg Lacosamide tablets taken for 50 -400 mg twice daily dosing for up to 2 years
  Other Names: Vimpat

SUMMARY:
This open-label extension trial will assess the long-term use of Lacosamide monotherapy and safety of Lacosamide monotherapy and adjunctive therapy in subjects with partial-onset seizures who were previously enrolled in the conversion to monotherapy trial (SP902).

ELIGIBILITY:
Inclusion Criteria:

* Subject has entered the Maintenance Phase of the double-blind trial, SP902, (ie, has taken at least 1 dose of SP902 Maintenance Phase trial medication) and either completed SP902 or met an exit criterion in SP902; subject is allowed up to 2 concomitant Antiepileptic Drugs (AEDs)

Exclusion Criteria:

* Subject meets the withdrawal criteria (excluding exit criteria) for the SP902 trial, or is experiencing an ongoing Serious Adverse Event (SAE)

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2008-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (108):
- United States (77):
  - 048, Alabaster, Alabama
  - 010, Birmingham, Alabama
  - 042, Northport, Alabama
  - 009, Phoenix, Arizona
  - 014, Phoenix, Arizona
  - 151, Phoenix, Arizona
  - 103, Tucson, Arizona
  - 102, Jonesboro, Arkansas
  - 007, Little Rock, Arkansas
  - 086, Little Rock, Arkansas
  - 120, La Habra, California
  - 059, Los Angeles, California
  - 021, Santa Monica, California
  - 107, Torrance, California
  - 060, Aurora, Colorado
  - 025, Fairfield, Connecticut
  - 094, Doral, Florida
  - 108, Gainesville, Florida
  - 123, Miami, Florida
  - 132, Miami, Florida
  - 077, Orlando, Florida
  - 049, Panama City, Florida
  - 129, Port Charlotte, Florida
  - 050, Sarasota, Florida
  - 004, Tallahassee, Florida
  - 079, Atlanta, Georgia
  - 058, Boise, Idaho
  - 131, Hines, Illinois
  - 146, Peoria, Illinois
  - 011, Springfield, Illinois
  - 078, Indianapolis, Indiana
  - 073, Ames, Iowa
  - 124, Manhattan, Kansas
  - 023, Wichita, Kansas
  - 160, Wichita, Kansas
  - 164, Lexington, Kentucky
  - 062, Louisville, Kentucky
  - 029, Scarborough, Maine
  - 020, Baltimore, Maryland
  - 034, Baltimore, Maryland
  - 065, Pikesville, Maryland
  - 137, Waldorf, Maryland
  - 041, Detroit, Michigan
  - 030, Golden Valley, Minnesota
  - 071, Hattiesburg, Mississippi
  - 031, Chesterfield, Missouri
  - 066, St Louis, Missouri
  - 017, Lebanon, New Hampshire
  - 067, Voorhees Township, New Jersey
  - 036, Albany, New York
  - 083, Buffalo, New York
  - 069, Cedarhurst, New York
  - 027, New York, New York
  - 122, New York, New York
  - 003, Asheville, North Carolina
  - 063, Durham, North Carolina
  - 117, Wilmington, North Carolina
  - 015, Cleveland, Ohio
  - 061, Columbus, Ohio
  - 002, Toledo, Ohio
  - 147, Oklahoma City, Oklahoma
  - 100, Greensburg, Pennsylvania
  - 032, Philadelphia, Pennsylvania
  - 024, Beaufort, South Carolina
  - 114, Chattanooga, Tennessee
  - 001, Nashville, Tennessee
  - 138, Austin, Texas
  - 022, Dallas, Texas
  - 046, El Paso, Texas
  - 051, Houston, Texas
  - 053, Houston, Texas
  - 098, San Antonio, Texas
  - 136, Layton, Utah
  - 161, Alexandria, Virginia
  - 016, Charlottesville, Virginia
  - 074, Renton, Washington
  - 080, Madison, Wisconsin
- Australia (5):
  - 421, Capmerdown, New South Wales
  - 425, Chatswood, New South Wales
  - 423, Herston, Queensland
  - 420, Adelaide, South Australia
  - 427, Parkville, Victoria
- Canada (7):
  - 140, Halifax, Nova Scotia
  - 116, Hamilton, Ontario
  - 093, London, Ontario
  - 091, Greenfield Park, Quebec
  - 110, Montreal, Quebec
  - 113, Montreal, Quebec
  - 127, Calgary
- 223, Aarhus, Denmark
- 461, Mainz, Germany
- Italy (3):
  - 443, Ferrara
  - 445, Reggio Calabria
  - 447, Torrette Di Ancona
- Poland (8):
  - 284, Częstochowa
  - 286, Gdansk
  - 282, Gdynia
  - 280, Krakow
  - 290, Lublin
  - 289, Szczecin
  - 281, Warsaw
  - 287, Warsaw
- 324, Santa Cruz de Tenerife, Spain
- United Kingdom (5):
  - 360, Blackpool
  - 367, Cornwall
  - 364, London
  - 369, London
  - 363, Middlesbrough

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Multicenter, Open-Label Study started to enroll Subjects in February 2008.
Pre-assignment Details: Participant Flow refers to the Safety Set, which is defined as all subjects who met the inclusion/exclusion criteria, signed an informed consent form, and took at least 1 dose of Trial medication.
Period: Overall Study
Arm/Group | Lacosamide
Started | 322
Completed | 210
Not Completed | 112
Not completed — Lack of Efficacy | 20
Not completed — Withdrawal by Subject | 30
Not completed — Fatal Serious AE | 3
Not completed — Non Fatal Serious AE | 7
Not completed — Non Fatal Non Serious AE | 12
Not completed — Protocol Violation | 3
Not completed — Unsatisfactory compliance of subject | 11
Not completed — Lost to Follow-up | 9
Not completed — Other reason for premature termination | 17

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set, which is defined as all subjects who met the inclusion/exclusion criteria, signed an informed consent form, and took at least 1 dose of Trial medication.
Arm/Group | Lacosamide
Number analyzed (Participants) | 322
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 301
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years]
  mean (standard deviation) | 40.7 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161
  Male | 161
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 258
  Black or African American | 46
  Asian | 1
  Other | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects on Lacosamide (LCM) Monotherapy at Any Time Between Visit 1 and End of Study
Description: Percentage of Subjects on Lacosamide (LCM) Monotherapy at any time between Visit 1 and End of Study.
Time Frame: From Visit 1 to End of Study (approximately 2 years)
Population: All 322 Subjects from the Safety Set are included in the Analysis of this Outcome Measure. Safety Set is defined as all subjects who met the inclusion/exclusion criteria, signed an informed consent form, and took at least 1 dose of Trial medication.
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 322
Participants | 292

2. Primary Outcome: Duration of Lacosamide (LCM) Monotherapy Treatment From Visit 1 to End of Study
Description: Duration of total Lacosamide Monotherapy From Visit 1 to End of Study.
Time Frame: From Visit 1 to End of Study (approximately 2 years)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Lacosamide
Number analyzed (Participants) | 322
days | 479.1 (271.9)

3. Secondary Outcome: Occurrence of At Least One Treatment-Emergent Adverse Event (TEAE) From Visit 1 to End of Study
Description: A TEAE is defined as any untoward medical occurrence (eg, noxious or pathological changes) in a subject or clinical investigation subject compared with pre-existing conditions, that occurs during any phase of a clinical trial including Pretreatment, Run-In, Wash-Out, or Follow-Up Phases.
  An TEAE is defined as being independent of assumption of any causality (eg, to trial or concomitant medication, primary or concomitant disease, or trial design).
Time Frame: From Visit 1 to End of Study (approximately 2 years)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 322
Participants | 296

4. Secondary Outcome: Occurrence of Treatment-Emergent Adverse Events (TEAE) Leading to Subject Withdrawal From Visit 1 to End of Study
Time Frame: From Visit 1 to End of Study (approximately 2 years)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 322
Participants | 22

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Study Start (Visit 1) until the End of Study (up to 2 years).
Description: Adverse Events refer to the Safety Set, which is defined as all subjects who met the inclusion/exclusion criteria, signed an informed consent form, and took at least 1 dose of Trial medication.
Arm/Group | Lacosamide
Serious Adverse Events (participants affected / at risk) | 56/322
Other Adverse Events (participants affected / at risk) | 238/322
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=322)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (2)
Sudden unexplained death in epilepsy (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (3)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Electroencephalogram (Investigations) | 1 (1)
Heart rate decreased (Investigations) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Convulsion (Nervous system disorders) | 17 (19)
Status epilepticus (Nervous system disorders) | 4 (6)
Syncope (Nervous system disorders) | 3 (3)
Postictal state (Nervous system disorders) | 2 (2)
Complicated migraine (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (2)
Migraine (Nervous system disorders) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Postictal psychosis (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=322)
Nausea (Gastrointestinal disorders) | 46 (68)
Vomiting (Gastrointestinal disorders) | 27 (37)
Diarrhoea (Gastrointestinal disorders) | 23 (27)
Fatigue (General disorders) | 40 (44)
Upper respiratory tract infection (Infections and infestations) | 45 (53)
Nasopharyngitis (Infections and infestations) | 38 (53)
Urinary tract infection (Infections and infestations) | 20 (30)
Influenza (Infections and infestations) | 19 (23)
Fall (Injury, poisoning and procedural complications) | 31 (44)
Contusion (Injury, poisoning and procedural complications) | 25 (49)
Laceration (Injury, poisoning and procedural complications) | 22 (32)
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 (41)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (18)
Dizziness (Nervous system disorders) | 89 (142)
Headache (Nervous system disorders) | 55 (81)
Convulsion (Nervous system disorders) | 29 (42)
Tremor (Nervous system disorders) | 26 (30)
Anxiety (Psychiatric disorders) | 24 (26)
Insomnia (Psychiatric disorders) | 20 (24)
Depression (Psychiatric disorders) | 17 (21)
Rash (Skin and subcutaneous tissue disorders) | 20 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days